CLINICAL TRIAL: NCT06720064
Title: Care Bundle Containing Chlorhexidine Dressing on Port Catheter and Central Venous Catheter-Related Bloodstream Infections in Pediatric Cancer Patients
Brief Title: Care Bundle Containing Chlorhexidine Dressing on Port Catheter and Central Venous Catheters
Acronym: CHG-port
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Afyonkarahisar Health Science University (Unknown)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: carebundle
Record Dates: First submitted 2024-09-18; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Cancer
Keywords: Care bundle; chlorhexidine; pediatric; cancer; catheter-related bloodstream infections
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care bundle approach; The following materials will be used by nurses while performing their care in accordance with the relevant care bundle and checklist;
  * Transparent catheter cover (3M™ IV-Tegaderm™) (Control group)
  * Needle-free interventional apparatus (BD Qsyte split septum™),
  * Prefilled flush syringe (BD PosiFlush™)
  * Alcohol swab (alcohol cloth),
  * Solupred Swab (3M™), (will be used to clean the dressing area)
- Care bundle approach with Chlorhexidine Dressing (Experimental): Care bundle approach with Chlorhexidine Dressing The following materials will be used by nurses while performing their care in accordance with the relevant care bundle and checklist;
  * Transparent catheter cover with Chlorhexidine (3M™ CHG Tegaderm™) (Study group)
  * Needle-free interventional apparatus (BD Qsyte split septum™),
  * Prefilled flush syringe (BD PosiFlush™)
  * Alcohol swab (alcohol cloth),
  * Solupred Swab (3M™), (will be used to clean the dressing area)
  Interventions: Device: Chlorhexidine Dressing

INTERVENTIONS:
Device: Chlorhexidine Dressing — Transparent catheter cover with Chlorhexidine (3M™ CHG Tegaderm™)
  Arms: Care bundle approach with Chlorhexidine Dressing

SUMMARY:
In order to provide treatment in pediatric hematology-oncology patients, in some cases a central venous catheter is required in children. The most important situation to pay attention to when using a central venous catheter is "Central line-associated bloodstream infections".

These infections are infections that develop after admission to the hospital and are not in the incubation period at the time of admission, or although they usually develop in the hospital 48-72 hours after hospitalization, they can sometimes appear after discharge. Central line-associated bloodstream infections significantly increase morbidity and mortality. In this context, the effect of using a care bundle containing chlorhexidine dressing on port catheter and central venous catheter-related bloodstream infections in pediatric cancer patients was examined.

DETAILED DESCRIPTION:
This study was designed as a prospective, cross-sectional, and randomized controlled study to examine the effect of a care package containing chlorhexidine dressing on port catheter and central venous catheter-related bloodstream infections in pediatric cancer patients.

Hypotheses of the Research H1: Care bundle approach including chlorhexidine dressing in pediatric cancer patients reduces port catheter and central venous catheter-related bloodstream infections.

H2: Care bundle approach including chlorhexidine dressing in pediatric cancer patients reduces port catheter and central venous catheter-related complications.

Randomization A stratified randomization scheme was used to distribute the sample into groups. Stratification randomization was made according to port catheter stay duration, age group, hematological/oncological cancer type and hematopoietic stem cell transplantation unit / pediatric hematology and oncology clinic.

ELIGIBILITY:
Inclusion Criteria:

* The child is receiving inpatient treatment at the Hematology and Oncology unit and hematopoietic stem cell transplantation unit
* The child has a diagnosis of hematological or oncological cancer
* The child's age range is between 1 and 17
* Having a port catheter inserted and no early complications have occurred
* The child agrees to participate in the study voluntarily
* The parent agrees to participate in the study voluntarily
* Obtaining the consent form from the child and parent
* He has been in the hospital for more than 48 hours

Exclusion Criteria:

* Have a systemic infection.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Central line-associated bloodstream infections | during the intervention, up to 1 years
  defined as the recovery of a pathogen from a blood culture in a patient who had a central line at the time of infection or within 48 hours before the development of infection

CONTACTS AND LOCATIONS:
Overall Officials: Gulcin Ozalp Gerceker, Assoc. Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No